CLINICAL TRIAL: NCT06231043
Title: Comparative Efficacy of Intramuscular Diclofenac Injection Versus Intravascular Tramadol Injection in Acute Renal Colic, a Randomized Controlled Trial
Brief Title: Diclofenac IM Versus Tramadol IV in Acute Renal Colic, RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lampang Hospital (Other)
Responsible Party: Principal Investigator, JARUPA YAOWALAORNG, JARUPA YAOWALAORNG, Lampang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100/66
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Acute Renal Colic
Keywords: Diclofenac IM versus Tramadol IV in acute renal colic, RCT
MeSH Terms: conditions — Renal Colic | interventions — Diclofenac; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug1 (Experimental): Diclofenac 75 mg (3 ml) IM injection by doctor, then followed by normal saline 20 ml IV injection (equal to Tramadol diluted) by nurse.
  Interventions: Drug: Diclofenac/Tramadol
- Drug2 (Active Comparator): Normal saline 3 ml IM injection by doctor (equal to Diclofenac 75 mg), then followed by Tramadol 50 mg (1 ml) dilute with normal saline 19 ml (total 20 ml )IV injection by nurse.
  Interventions: Drug: Diclofenac/Tramadol

INTERVENTIONS:
Drug: Diclofenac/Tramadol — Arm Drug1 :Diclofenac 75 mg (3 ml) IM injection by doctor, then followed by normal saline 20 ml IV injection (equal to Tramadol diluted) by nurse.
  Arm Drug2 :Normal saline 3 ml IM injection by doctor (equal to Diclofenac 75 mg), then followed by Tramadol 50 mg (1 ml) dilute with normal saline 19 ml (total 20 ml )IV injection by nurse.
  Other Names: Fenac/Tramol

SUMMARY:
Patients presented with acute pain from renal colic, the standard of care are prescribed NSAIDs, most common drug used is intramuscular (IM) Diclofenac injected at the gluteal muscle. Due to adverse effects in some patients, the nursing council has banned the injection by nurses. Since then, there has been a change in treatment by using intravascular (IV) Tramadol. According to various research, Diclofenac has a higher efficacy in controlling pain compared to other medications. In clinical practice, Tramadol has less efficacy of decreasing pain and a longer onset of action. At presence, there has been no research performed comparing the efficacy between these two drugs especially from the viewpoint of time dimension.

DETAILED DESCRIPTION:
To compare the efficacy Diclofenac 75 mg IM versus Tramadol 50 mg IV in patients with acute pain from renal colic.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Acute pain in renal/ureteric colic
3. Pain score more than 4
4. Confirmation diagnosis by ultrasound bedside

Exclusion Criteria:

1. Refused to participate in the research
2. Pregnancy
3. Contraindicated of Diclofenac or Tramadol
4. Urinary tract infection
5. Skin infection at Buttock area
6. Acute kidney injury
7. CKD stage III, IV, V
8. Bilateral severe hydronephrosis
9. Physician refusal

Min Age: 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Diclofenac 75 mg IM or Tramadol 50 mg IV | 30,60,90,120 minutes
  Time to pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Jarupa Yaowalaorng, Principal Investigator — Lampang Hospital
Locations (1):
- Lampang hospital, Lampang, Thailand

IPD SHARING:
Plan to Share IPD: No
Personal reasons